CLINICAL TRIAL: NCT05297734
Title: Comparative Effectiveness Trial of Two Supportive Cancer Care Delivery Models for Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 63646
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: End of Life; Cancer
Keywords: Carcinoma; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Pancreatic Neoplasms; Sarcoma; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Stomach Neoplasms; Glioblastoma; Rectal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Breast Neoplasms; Carcinoma, Renal Cell; Skin Neoplasms; Small Cell Lung Carcinoma; Osteosarcoma; Myelodysplastic Syndromes; Disease Progression; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Urogenital Neoplasms; Carcinoma, Bronchogenic
MeSH Terms: conditions — Death; Neoplasms; Carcinoma; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Pancreatic Neoplasms; Sarcoma; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Stomach Neoplasms; Glioblastoma; Rectal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Breast Neoplasms; Carcinoma, Renal Cell; Skin Neoplasms; Small Cell Lung Carcinoma; Osteosarcoma; Myelodysplastic Syndromes; Disease Progression; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Urogenital Neoplasms; Carcinoma, Bronchogenic

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial among 26 clinics
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-based supportive cancer care (Active Comparator): Patients receive educational materials to assist with advance care planning and symptom management through a technology-based supportive cancer care weekly during months 1-4 and every other week during months 5-12.
  Interventions: Other: Receive technology-based supportive cancer care
- Redesigned team-based supportive cancer care (Experimental): Patients are paired with a health educator who will discuss the same educational materials from ARM A either in person or by telephone discussions weekly during months 1-4 and every other week during months 5-12.
  Interventions: Behavioral: Receive redesigned team-based supportive cancer care

INTERVENTIONS:
Other: Receive technology-based supportive cancer care — All participants will receive an electronic health record message or email with standardized information provided regarding advance care planning and symptom management.
  Other Names: Technology-based SCC approach
  Arms: Technology-based supportive cancer care
Behavioral: Receive redesigned team-based supportive cancer care — Lay Health Workers will meet with 1:1 with participants over 12 months to discuss advance care planning, surrogate decision-makers, advance directives and physician orders for life sustaining treatment.
  Other Names: Patients Activated in Cancer care through Teams (PACT), Redesigned SCC team-based approach
  Arms: Redesigned team-based supportive cancer care

SUMMARY:
This cluster-randomized comparative effectiveness trial compares a technology-based supportive cancer care (SCC) approach with a redesigned team-based supportive cancer care (SCC) approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Greater intervention effects on health-related quality of life

SECONDARY OBJECTIVES:

I. Greater intervention effects on patient activation II. Greater satisfaction with care and decision-making III. Greater documentation of goals of care and symptoms IV. To lower acute care V. Greater palliative care and hospice

OUTLINE: Sites are randomized to 1 of 2 arms.

ARM A: Patients receive educational materials to assist with advance care planning and symptom management through a technology-based supportive cancer care weekly during months 1-4 and every other week during months 5-12.

ARM B: Patients are paired with a lay health worker who will discuss the same educational materials from ARM A either in person or by telephone discussions weekly during months 1-4 and every other week during months 5-12.

All participants complete a baseline interview upon enrollment during the initial consent phone contact and then a survey at 3-, 6-and 12-months post enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with solid tumor cancer diagnosis or recurrence of the disease.
2. Patients must have the ability to understand and willingness to provide verbal consent.
3. Participants must speak English, Spanish, Chinese, or Vietnamese.

Exclusion Criteria:

1. Inability to consent to the study
2. Plans to change oncologist within 12 months
3. Employed by the practice site
4. Patients who anticipate moving from the area within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2996 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life as assessed by the Functional Assessment of Cancer Therapy (FACT-G). | Change in health-related quality of life from baseline to 3 months
  Each patient will receive a health-related quality of life survey (FACT-G) at baseline, 3 months, 6 months, and 12 months.

SECONDARY OUTCOMES:
Change in health-related quality of life as assessed by the Functional Assessment of Cancer Therapy (FACT-G). | Change in health-related quality of life from baseline to 6, and 12 months
  Each patient will receive a health-related quality of life survey (FACT-G) at baseline, 3 months, 6 months, and 12 months.
Change in patient activation using the Patient Activation Measure (PAM-13). | Change in patient activation from baseline to 3, 6, and 12 months
  Each patient will receive a validated patient activation survey (PAM-13) to assess their activation at baseline, 3 months, 6 months, and 12 months.
Change in satisfaction with care using the Consumer Assessment of Health Care (Providers and Systems (CAHPS) Cancer Care Survey Questions #39 and #42. | Change in satisfaction with care from baseline to 3, 6, and 12 months
  Each patient will receive a validated satisfaction with care survey at baseline, 3 months, 6 months, and 12 months.
Change in satisfaction with decision using the Satisfaction with Decision Scale (SWD) | Change in satisfaction with decision from baseline to 3, 6, and 12 months
  Each patient will receive a validated satisfaction with decision survey at baseline, 3 months, 6 months and 12 months.
Palliative Care Use (Self-reported and Chart Review) | 3, 6, and 12 months after patient enrollment
  Palliative care use will be self-reported by each patient or abstracted by electronic medical record at 3, 6 and 12 months after patient enrollment.
Hospice Care Use (Self-reported and Chart Review) | 3, 6, and 12 months after patient enrollment
  Hospice care use will be self-reported by each patient or abstracted by electronic medical record at 3, 6, and 12 months after patient enrollment.
Emergency Department Visits (Self-reported and Chart Review) | 3, 6, and 12 months after patient enrollment
  Emergency Department use will be self-reported by each patient or abstracted by electronic medical record at 3, 6, and 12 months after enrollment.
Hospitalization Visits (Self-reported and Chart Review) | 3, 6, and 12 months after patient enrollment
  Hospital use for each patient will be self-reported by each patient or abstracted by electronic medical record at 3, 6, and 12 months after enrollment.
Documentation of goals of care discussions (Chart Review) | 3, 6, and 12 months after patient enrollment
  Documentation of goals of care discussions will be abstracted by electronic medical record chart review for each patient at 3, 6, and 12 months after enrollment.
Documentation of symptom discussions (Chart Review) | 3, 6, and 12 months after patient enrollment
  Documentation of symptom discussions will be abstracted by electronic medical record chart review for each patient at 3, 6, and 12 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Beckman Research Institute of City of Hope, Duarte, California
  - VA Medical Center, Fresno, Fresno, California
  - Santa Clara Valley Medical Center, Fruitdale, California
  - St Jude Heritage Medical Group, Fullerton, California
  - Oncology Institute for Hope and Innovation, Los Angeles, California
  - Sacramento VA Medical Center - VA Northern California Health Care System, Mather, California
  - Pacific Cancer Care, Monterey, California
  - VA Palo Alto, Palo Alto, California
  - Zuckerberg San Francisco General, San Francisco, California
  - Kaiser Foundation Research Institute, San Francisco, California
  - University of San Francisco, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - Spark M. Matsunaga VA Medical Center, Honolulu, Hawaii
  - North Las Vegas VA Medical Center, Las Vegas, Nevada
  - George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah